CLINICAL TRIAL: NCT05056740
Title: Evaluation of a Combined Analysis of Serum and Cerebrospinal Fluid Inflammatory Biomarkers to Help in Etiological Diagnosis of Central Nervous System Autoimmune Diseases
Brief Title: Combined Analysis of Inflammatory Biomarkers for CNS Autoimmune Diseases Diagnostic
Acronym: CyBIRD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Neuro02
Record Dates: First submitted 2021-09-16; First posted 2021-09-24 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Central Nervous System Diseases
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MS: Patients with a definite MS diagnosis according to the 2017 McDonald criteria
  Interventions: Biological: Data analysis
- Red-flag MS: Patients presenting with clinical, radiological or biological red flags for MS diagnosis who will be ultimately diagnosed as having MS
  Interventions: Biological: Data analysis
- Other CNS autoimmune diseases: Patients with a definite diagnostic of CNS autoimmune disease that is not MS
  Interventions: Biological: Data analysis
- Controls: Patients with a definite diagnostic of non-inflammatory CNS disorder
  Interventions: Biological: Data analysis

INTERVENTIONS:
Biological: Data analysis — Analysis of the data from routine care at the end of the diagnostic work-up

SUMMARY:
Project rationale:

Since 2017, multiple sclerosis diagnosis should match the new McDonald criteria in which a "no better explanation than MS" should be fulfilled. However, many patients present with red flags that lead to a complex diagnostic work-up. There are no available biomarkers that permit to confirm or roll out MS diagnosis in such cases. Therefore, we lack biological markers that can help in the diagnosis of patients presenting with suspected MS.

Many studies have found that serum and cerebrospinal fluid (CSF) cytokines could help to differentiate MS from other diseases such as neuromyelitis optica spectrum disorders (i.e., IL-6) or neurosarcoidosis (i.e., sIL-2R). Serum and CSF kappa free light chains have also shown good diagnosis performance in MS. In daily practice, our MS tertiary center already perform the analysis of CSF concentrations of IL-1β, sIL-2R, IL-6, IL-10, and serum and CSF kappa and lambda free light chains to roll out other central nervous system (CNS) autoimmune diseases in patients presenting with white matter hyperintensities (WMH).

Objective:

To correlate CSF IL-1β, sIL-2R, IL-6, IL-10, serum and CSF kappa and lambda free light chains with the final diagnosis in patients presenting to our MS tertiary center with suspected MS to identify a specific inflammatory biomarker profil involved in MS and other CNS autoimmune diseases.

The methodology:

This is an observational study. All patients ongoing a routine diagnostic work-up for suspected MS from june 2020 to june 2022 in our MS tertiary center will be analyzed. Cerebrospinal fluid IL-1β, sIL-2R, IL-6, IL-10, serum and CSF kappa and lambda free light chains will be correlated with the final diagnosis to ultimately find MS associated biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our center for the diagnostic work-up of White Matter Lesions
* Patients that need a routine blood analysis
* Patients that need a routine CSF analysis
* Non opposition to research consent

Exclusion Criteria:

* Patients with a contraindication to perform spinal tap (increase bleeding risk medicine or disease)
* Patients with a contraindication to MRI (metal prosthesis…)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred to our MS tertiary center for the diagnostic work-up of white matter hyperintensities suggestive of underlying inflammatory demyelinating disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Identify specific biomarkers profil in MS group | 1 day
  Quantification in each group of patients of IL-1beta, soluble receptor of IL-2, IL-6 and IL-10 by ELISA and cerebrospinal fluid/serum kappa and lambda free light chains by using the turbidimetric analyzer Optilite (BindingSite).

SECONDARY OUTCOMES:
To define the diagnosis performance of "Central vein sign (CVS)" in Radiologically Isolated Syndrome subjects compared to MS patients and patients with WM abnormalities of another origin. | 1 day
  Proportion of CVS positive lesions in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided